CLINICAL TRIAL: NCT04355793
Title: An Open-Label Expanded Access Program of Ruxolitinib for the Emergency Treatment of Cytokine Storm From COVID-19 Infection
Brief Title: Expanded Access Program of Ruxolitinib for the Emergency Treatment of Cytokine Storm From COVID-19 Infection
Status: No longer available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: INCB 18424-MA-COVID-19-301
Record Dates: First submitted 2020-04-18; First posted 2020-04-21 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Cytokine Storm; ruxolitinib
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — ruxolitinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib starting dose level 5 mg orally, twice daily (BID).
  Other Names: INCB018424

SUMMARY:
To provide ruxolitinib through an expanded access program for the treatment of cytokine storm due to COVID-19 in the United States to patients who are eligible but not able to be hospitalized or who are hospitalized with a clinical diagnosis and/or positive test for SARD-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 12 years of age or older.
* Clinical diagnosis of COVID-19 and/or locally accepted positive test; if feasible, swab should be taken and saved for quantitative testing to determine viral load.
* Disease severity making the patient eligible for hospitalization (whether or not hospitalization is available), with evidence of cytokine storm as determined by the treating physician. Manifestations of cytokine storm can include the following:
* Severe shortness of breath (respiratory rate > 24 breaths/minute).
* SpO2 of < 90% on ambient air.
* Need for invasive or noninvasive mechanical ventilation.
* Acute respiratory distress syndrome.
* Multiple organ failure.
* Be willing to avoid pregnancy or fathering children
* Able to provide written informed consent, consent from the patient's legally authorized representative, and/or assent from the patient, parent, or guardian.

Exclusion Criteria:

* Patients, patient's legally authorized representative, or legal guardians unable to review and sign ICF.
* Females who are pregnant or breastfeeding, and males and females who cannot comply with requirements to avoid fathering a child or becoming pregnant.
* Patients with inadequate liver function (ALT above 4 × ULN or direct bilirubin 4 × ULN and the laboratory abnormalities are considered to be due to underlying liver dysfunction).
* Patients with platelet counts < 50 × 109 /L
* Any underlying or current medical or psychiatric condition that, in the opinion of the treating physician, would place the patient at an unacceptable risk if he or she were to participate in the program.
* Previous allergic reactions to JAK inhibitors or excipients.
* Concomitant use of any other JAK inhibitor.
* Is eligible or able to access ruxolitinib through an Incyte-sponsored clinical study or is eligible for another therapeutic clinical trial for cytokine storm at the treating institution..

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] Weinstein J, Jagan N, Lorthridge-Jackson S, Hamer-Maansson JE, Squier P. Ruxolitinib for Emergency Treatment of COVID-19-Associated Cytokine Storm: Findings From an Expanded Access Study. Clin Respir J. 2025 Apr;19(4):e70050. doi: 10.1111/crj.70050. PMID 40197709